CLINICAL TRIAL: NCT06751394
Title: Preoperative Treatment with Radiotherapy and Anti-PD1 for Resectable Recurrent Rectal Cancer (TRACER)
Brief Title: Preoperative Chemoradiotherapy and Toripalimab in Locally Recurrent Rectal Cancer
Acronym: TRACER
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiaojian Wu, hospital director, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024ZSLYEC-684
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Recurrent Rectal Cancer
Keywords: locally recurrent rectal cancer; PD-1 inhibitor; preoperative chemoradiotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — toripalimab; Capecitabine; Oxaliplatin; Irinotecan; Radiation; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Group A (Experimental): The patients will receive 2 cycles of XELOX or XELIRI and PD-1 antibody, followed by long course radiotherapy (45-50Gy/25f or 30Gy/25f), concurrent with Capecitabine and 1-2 cycles of PD-1 antibody, then receive 2-3 cycles of XELOX or XELIRI and PD-1 antibody. Curative surgery is scheduled after neoadjuvant treatment.
  Interventions: Drug: PD-1 antibody (Toripalimab); Drug: Capecitabine; Drug: Oxaliplatin; Drug: Irinotecan; Radiation: Radiation; Procedure: surgery

INTERVENTIONS:
Drug: PD-1 antibody (Toripalimab) — PD-1 antibody: (Toripalimab): 240mg q3w
Drug: Capecitabine — Capecitabine:1000mg/m² d1-14 q3w; Capecitabine:825mg/m² on the day of radiotherapy
Drug: Oxaliplatin — 130 mg/m² q3w
Drug: Irinotecan — 200 mg/m² q3w
Radiation: Radiation — 45-50Gy/25Fx or 30Gy/15Fx
Procedure: surgery — The type of surgery will depend on the site of recurrence and the involvement of adjacent structures, which will be determined by the surgeons.

SUMMARY:
The study is a prospective, single-center, single-arm, phase II clinical trial. Patients with pelvic recurrent rectal cancer aged from 18 to 75 years, Eastern Cooperative Oncology Group performance status of 0-1, will receive 45-50Gy/25Fx irradiation or 30Gy/15Fx reirradiation (history of pelvic radiation). PD-1 inhibitor (Toripalimab) was used throughout the course of induction chemotherapy (before radiation), concurrent chemoradiation and consolidation chemotherapy (after radiation); radical resection was followed by well-experienced surgeons .

The primary endpoint was pathological complete response (pCR) rate. Secondary endpoints were R0 resection rate, 3-year progression-free survival, overall survival, pathological tumor regression grade, operation characteristics and incidence of major surgical complications.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 18-75 years old at the time of signing the informed consent form.
2. ECOG performance status 0-1.
3. Pathological confirmed or MRI/ enhanced CT confirmed pelvic recurrence.
4. No distant metastasis lesions outside the pelvic.
5. No prior radiotherapy within 6 months.
6. Participants with pelvic recurrence who have not previously been treated with first-line chemotherapy.
7. Life expectancy at least 24 weeks.
8. Adequate organ function (bone marrow, liver, kidney and clotting function) within 7 days before the first administration without using blood products or hematopoietic stimulating factors.
9. Non pregnancy or lactation.
10. Fully informed and willing to provide written informed consent for the trial.

Exclusion Criteria:

1. Neutrophil < 1.5×10^9/L, PLT < 75×10^9/L.
2. TBIL > 1.5 ULN.
3. AST or ALT > 2.5 ULN, or ALT and / or AST > 5 ULN in patients with liver metastasis.
4. Cr > 1.5 ULN.
5. Serious electrolyte abnormalities.
6. Active coronary artery disease, severe/unstable angina, or newly diagnosed angina or myocardial infarction within 12 months.
7. Arterial thrombosis or deep vein thrombosis within 6 months, such as cerebrovascular accidents (including transient ischemic attacks), pulmonary embolism, deep vein thrombosis.
8. Congestive cardiac failure ≥ NYHA grade 2.
9. Human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS), untreated active hepatitis (hepatitis B defined as HBV-DNA ≥ 500 IU/ml; hepatitis C defined as HCV-RNA higher than lower limit of detection) or hepatitis B and hepatitis C virus co-infection.
10. Active inflammatory bowel disease or other colorectal diseases that lead to chronic diarrhea.
11. Suspected autoimmune disease.
12. Interstitial lung disease, non-infectious pneumonia or uncontrollable systemic diseases (such as diabetes, hypertension, pulmonary fibrosis and acute pneumonia).
13. Suspected allergic to any drugs used in the trial.
14. History of any immune checkpoint inhibitor therapy.
15. Clinically detectable second primary malignancy, or history of other malignancies within 5 years.
16. Pregnant or lactating women or women who may be pregnant have a positive pregnancy test before the first medication; Or the female participants themselves and their partners who were unwilling to implement strict contraception during the study period.
17. The investigator considers that the subject is not suitable to participate in this clinical study due to any clinical or laboratory abnormalities or compliance problems.
18. Serious mental abnormalities.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate | up to 1 year
  Defined as pathological evaluation of resected tumor tissue and regional lymph nodes, with no residual tumor cells, complete disappearance of all tumor lesions, and no appearance of new lesions.

SECONDARY OUTCOMES:
R0 resection rate | up to 1 year
  Complete resection rate, defined as no residual tumor cells at the surgical margin under the microscope or the naked eye.
3-year Progression-Free Survival | up to 3 years
  Defined as the time from the date of start treatment until the date of local recurrence or local recurrence progression or distant metastases or death from any cause or censored at last follow-up within 3 years.
Overall Survival | up to 3 years
  Defined as the time from the date of start treatment until the date of death from any cause or censored at last follow-up.
Pathological tumor regression grading | up to 1 year
  Classify according to the Mandard tumor regression grading system.
Operation complications | up to 1 year
  intraoperative complications
Incidence of major surgical complications | up to 3 months
  From the date of surgery to 3 months after surgery, according to Clavien-Dindo classification score.

CONTACTS AND LOCATIONS:
Locations (1):
- Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided